CLINICAL TRIAL: NCT02056145
Title: Ultrasound Guided Lateral Femoral Cutaneous Block (LFCNB) And Femoral Nerve Block (FNB) For Postoperative Pain Control After Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Ethische Comité UZ Antwerpen, University Hospital, Antwerp
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/36/241
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: -Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Placebo Comparator): Group 1 consented subjects who will receive for their hip surgery procedures general anesthesia (sevoflurane) with single shot femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 cc of 0.9% saline solution for the femoral block and 10 cc of 0.9% saline solution for lateral femoral cutaneous block, for a total of 30 ml saline solution 0.9%.
  Interventions: Procedure: LFCNB; Procedure: FNB
- Group 2 (Active Comparator): Group 2 consented subjects who will receive for their hip surgery procedures general anesthesia (sevoflurane) with single shot femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 cc of 0.25% bupivacaine solution for the femoral block and 10 cc of 0.9% saline solution for lateral femoral cutaneous block, for a total of 20 cc 0.25% bupivacaine solution en 10 cc saline solution 0.9%.
  Interventions: Procedure: LFCNB; Procedure: FNB
- Group 3 (Active Comparator): Group 3 consented subjects who will receive for their hip surgery procedures general anesthesia (sevoflurane) with single shot femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 cc of 0.25% bupivacaine solution for the femoral block and 10 cc of 0.25% bupivacaine solution for lateral femoral cutaneous block, for a total of 30 cc of 0.25% bupivacaine solution.
  Interventions: Procedure: LFCNB; Procedure: FNB

INTERVENTIONS:
Procedure: LFCNB — LFCNB - Normal Saline solution 10 cc
  Arms: Group 1; Group 2
Procedure: FNB — FNB - Normal saline solution 10 cc
  Arms: Group 1
Procedure: LFCNB — LFCNB - Chirocaine 0.25%, 20 cc
  Arms: Group 3
Procedure: FNB — FNB - Chirocaine 0.25%, 20 cc
  Arms: Group 2; Group 3

SUMMARY:
Evaluation of the combination of lateral femoral cutaneous nerve "single shot" and femoral nerve "single shot" block as effective and safe alternative postoperative analgesic technique after hip replacement surgery.

DETAILED DESCRIPTION:
Clinical evaluation via a prospective, double-blinded, randomized clinical trial, whether ultrasound-guided single femoral block and lateral femoral cutaneous nerve blocks with 20 en 10 cc bupivacaine 0.25% respectively vs. the only ultrasound-guided single femoral block with 20 cc bupivacaine 0.25%, given just prior to elective hip surgery procedure, is effective in reducing acute postoperative pain (VAS scores) and postoperative opiate consumption.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip arthroplasty with posterolateral approach.

Exclusion Criteria:

* Known allergy to levobupivacaine and / or piritramide
* Known neurological disorders or peripheral neuropathies
* Existing drug or alcohol abuse
* Chronic use of pain medication (> started 3 months ago) not related to the hip suffering
* Coagulopathy (international normalized ratio) > 1.4
* Thrombocytopenia <70,000 platelets,
* Dementia
* Pregnancy
* Local infection hip
* Hepatic and / or renal impairment
* BMI> 45.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Use of opioids | 48 hours
  The primary outcome measure will be a consumption of opioids through the Intravenous Patient Controlled Analgesia pump. Those amounts will be measured en documented at the fixed intervals during the first 48 hours post-procedure.

SECONDARY OUTCOMES:
Visual analog scale (VAS) scores (0-10) | 48 hours
  The secondary outcome measure will be pain scores (VAS 0-10). Those scores will be measured en documented at the fixed intervals during the first 48 hours post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan TEMURZIEV, MD, Principal Investigator — Department of Anesthesiology, Antwerp University Hospital
Locations (1):
- AZ Sint Augustinus, Wilrijk, Antwerpen, Belgium